CLINICAL TRIAL: NCT01558037
Title: A Study to Correlate CMV-Specific Cell Mediated Immunity With Risk of CMV Disease and With Clinical Response to Therapy Following Solid Organ Transplantation
Brief Title: Cell Mediated Immunity With Risk of Cytomegalovirus (CMV) in Solid Organ Transplant Recipients
Acronym: ViracorCMI
Status: Completed | Type: Observational
Sponsor: Michael Ison (Other)
Collaborators: ViraCor Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Michael Ison, Associate Professor, Northwestern University
Organization: Northwestern University (Other)
Other Study IDs: NU-ViraCor 001
Record Dates: First submitted 2012-03-14; First posted 2012-03-20 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Awaiting Organ Transplant; Infection in Solid Organ Transplant Recipients
Keywords: transplant; solid organ transplant; kidney transplant; liver transplant; pancreas transplant; heart transplant; CMV; Cytomegalovirus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Main study: Main study patients are enrolled before or at time of solid organ transplant. Qualifying subjects either have tested positive for Cytomegalovirus or have a donor who has tested positive for Cytomegalovirus.
- Sub study: Subjects are enrolled to this arm who have begun replicating Cytomegalovirus post transplant. These subjects may or may not have been on the main study arm.

SUMMARY:
Cytomegalovirus (CMV) is a common infection with 60-90% of all adults worldwide having evidence of having the infection at sometime in their life. Patients who have undergone transplantation are at risk at developing CMV, especially those patients who do not have antibodies to CMV pre-transplant, but received an organ from a recipient who has antibodies to CMV. Usually the disease CMV causes is mild and sometimes patients are not even aware they have the infection without tests to detect the virus. CMV can less commonly cause serious infections that affect many parts of the body including the intestines, liver, or lungs. In rare cases CMV infection in transplant patients can cause death.

All patients who receive a transplant are monitored for CMV infection. The purpose of this study is to determine if there is a way the investigators can determine in advance which patients are at greatest risk of CMV infection. Specifically, this study will analyze the immune system of transplant patients to determine if there are specific elements of the immune system that 1) helps protect the body against CMV infection, and 2) helps the body combat CMV once it is infected. Identifying these specific elements of the immune system could improve the physician's ability to monitor the SOT patients for CMV infection, and to help treat CMV in those patients that become infected.

DETAILED DESCRIPTION:
Our hypothesis is that the degree of CMV cell-mediated immune (CMI) response correlates inversely with the risk of development of CMV replication and correlates with the response to initial therapy and risk of relapse after onset of replication. The primary aim of this study is to determine an association between CMV CMI response and both the risk of CMV infection and the degree of initial CMV viremia and rate of viremia clearance with standard CMV therapy. The first secondary aim is to determine an association between CMV QnPCR, CMV microRNA expression, TLR2 expression, and CMV-specific CMI and the risk of relapse of CMV disease after initial treatment. The second secondary aim is to determine an association between CMV QnPCR, CMV microRNA expression, TLR2 expression, and CMV-specific CMI collected at CMV infection and the following prospective data: Development of CMV end organ disease, resolution of symptoms of CMV infection, other non-CMV infections after initial CMV infection, graft rejection, recurrent or resistant CMV infection, and other markers of immune function. The third secondary aim is to determine an association between CMV QnPCR, CMV microRNA expression, TLR2 expression, and CMV-specific CMI response collected at CMV infection in solid-organ transplant (SOT) recipients and the following retrospective data: Type of SOT, CMV donor/recipient status, type and degree of immunosuppression, type and length of CMV prophylaxis, prior graft rejection and infections (non-CMV).

ELIGIBILITY:
Inclusion Criteria:

* Main Study Subjects will be recruited if they are listed for a SOT (liver, liver-kidney, kidney, kidney-pancreas, cardiac). At the time of transplant, consented patients will have an immediate pre-transplant blood draw for baseline labs subsequent labs will only be drawn if the donor/recipient CMV serostatus is CMV D+/R- (up to a maximum of 50 subjects) or D+/R+ or D-/R+ (up to a maximum of 50 subjects). Subjects must be ≥ 18 years of age, be consentable, and agree to have laboratory and clinical follow-up at Northwestern.
* CMV Replication Substudy
* Subjects will be recruited if they have undergone SOT, are found to have a positive CMV QnPCR (> 600 copies/mL) and will be subsequently treated for CMV infection with either intravenous ganciclovir or oral valganciclovir therapy at the discretion of the treating provider. Subjects must be ≥ 18 years of age, able to give consent, and agree to have laboratory and clinical follow-up at Northwestern.

Exclusion Criteria:

* Subjects will be excluded if they have had a previous history of CMV infection after SOT prior to enrollment (a prior episode of CMV infection or replication prior to the onset of the current episode). Subjects will also be excluded if the subject cannot give informed consent or if the subject is not able to comply with follow-up testing and/or treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The main study will recruit adult solid organ transplant recipients at Northwestern Memorial Hospital who are CMV donor positive, recipient negative (D+/R-) and SOT recipients at NMH who are CMV recipient positive, irrespective of donor status (D±/R+). A sub-study of this study will enroll up to 50 adult SOT recipients who have quantifiable CMV DNA by PCR and require CMV antiviral therapy, irrespective of their participation in the main study. Patients will be identified prior to transplantation as part of the pre-transplant evaluation process and will be consented either pre-transplant or on the first post-operative day in which they can provide written consent.
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Assessment of CMV Cell-Mediated Immune Response | For 8 months after transplant or 4 months after clearance of CMV
  Association between CMV CMI response and both the risk of CMV infection and the degree of initial CMV viremia and rate of viremia clearance with standard CMV therapy

SECONDARY OUTCOMES:
Assessment of CMV QnPCR, CMV microRNA expression, TLR2 expression, and CMV-specific CMI | For 8 months after transplant or 4 months after clearance of CMV
  Association between CMV QnPCR, CMV microRNA expression, TLR2 expression, and CMV-specific CMI collected at CMV infection and the following prospective data:
  * Development of CMV end organ disease
  * Resolution of symptoms of CMV infection
  * Other non-CMV infections after initial CMV infection
  * Graft rejection
  * Recurrent or resistant CMV infection
  * Other markers of immune function
  * Type of SOT
  * CMV donor/recipient status
  * Type and degree of immunosuppression
  * Type and length of CMV prophylaxis
  * Prior graft rejection and infections (non-CMV)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Ison, MD,MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States